CLINICAL TRIAL: NCT03760484
Title: Serial Fecal Microbiota Transplant (FMT) Plus Fidaxomicin in the Treatment of Severe or Fulminant Clostridium Difficile Infection, With Detailed Characterization in Microbiota, Metabolomics and Host Immune Response
Brief Title: Fecal Microbiota Transplant (FMT) Plus Fidaxomicin for Severe or Fulminant Clostridium Difficile Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty enrolling participants/COVID pandemic/lack of continued in-kind support from product manufacturer.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00081229
Record Dates: First submitted 2018-11-15; First posted 2018-11-30 (Actual); Results first posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-10

CONDITIONS: Clostridium Difficile
Keywords: Fecal microbiota transplantation; Fidaxomicin
MeSH Terms: interventions — Fidaxomicin; Fecal Microbiota Transplantation; Biological Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- fecal transplant with fidaxomicin (Experimental): FMT per rectum x 3 days in conjunction with fidaxomicin (dificid) PO 200 mg bid x 7-10 days
  Interventions: Drug: Fidaxomicin 200 mg; Biological: fecal microbiota transplantation (FMT)

INTERVENTIONS:
Drug: Fidaxomicin 200 mg — Each cycle consists of fidaxomicin 200 mg PO bid x 7-10 days till clinical efficacy is achieved, to a max of 4 cycles.
  Other Names: dificid
Biological: fecal microbiota transplantation (FMT) — Each cycle consists of FMT per rectum daily x 3 days till clinical efficacy is achieved to a max of 4 cycles
  Other Names: biotherapy

SUMMARY:
Fecal microbiota transplantation (FMT) has been very effective for patients who suffer from mild C diff infection (CDI) which recurs but it is unclear how effective FMT alone is in treating severe and fulminant CDI. Current evidence suggests that FMT in combination with vancomycin is required, and that multiple treatments are necessary. The investigators think fidaxomicin may be a better option in the context and may potentially reduce the number of FMT required. However, fidaxomicin has never been used to treat severe or fulminant CDI. In this pilot study, the investigators plan to use a combination of FMT plus fidaxomicin to determine efficacy and safety in treating patients with severe or fulminant CDI. The investigators want to see if this approach may reduce the number of FMT treatment required, and/or the length of hospital stay.

DETAILED DESCRIPTION:
In this prospective, open -label, multi--center feasibility study, the investigators aim to determine the efficacy and safety of using combined serial FMT by enema plus fidaxomicin to treat patients who have severe or fulminant CDI not responding to maximal medical therapy. The hypothesis is the combination of FMT plus fidaxomicin can reduce the number of FMT required and/or hospital length of stay compared to FMT plus vancomycin.

Participants will receive FMT by enemas over 3 days which constitutes a single cycle with concurrent treatment with oral fidaxomicin. If participants do not show improvement biochemically or clinically, then a repeat FMT cycle will be administered to a maximum of 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years with severe1 or fulminant2 CDI, without an adequate response to metronidazole IV 500 mg q8H and vancomycin 500 mg PO q6h for at least 2 days or after Fecal Microbiota Transplant (FMT). An adequate response is defined as a decrease in stool frequency or inflammatory markers (WBC or C reactive protein) by 10% over 48 hours
* Those with ability to provide informed consent or an alternative decision maker providing assent

Exclusion Criteria:

* Those with bowel perforation
* Those taking chemotherapy or radiation treatment with absolute neutrophil count of < 1000 cells/mm3
* Those with known colonic strictures
* Those with subtotal colectomy or planning to have a colectomy
* Those with significant ileus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Kao, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monaghan TM, Duggal NA, Rosati E, Griffin R, Hughes J, Roach B, Yang DY, Wang C, Wong K, Saxinger L, Pucic-Bakovic M, Vuckovic F, Klicek F, Lauc G, Tighe P, Mullish BH, Blanco JM, McDonald JAK, Marchesi JR, Xue N, Dottorini T, Acharjee A, Franke A, Li Y, Wong GK, Polytarchou C, Yau TO, Christodoulou N, Hatziapostolou M, Wang M, Russell LA, Kao DH. A Multi-Factorial Observational Study on Sequential Fecal Microbiota Transplant in Patients with Medically Refractory Clostridioides difficile Infection. Cells. 2021 Nov 19;10(11):3234. doi: 10.3390/cells10113234. PMID 34831456

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fecal Transplant With Fidaxomicin
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fecal Transplant With Fidaxomicin
Number analyzed (Participants) | 4
Age, Customized [Count of Participants; unit: Participants]
  60-69 years | 1
  70-79 years | 1
  80+ years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 4

OUTCOME MEASURES:

1. Primary Outcome: C Difficile Infection (CDI) Resolution- Short Term (Two Weeks After Final Fecal Microbiota Transplant (FMT))
Description: Defined as <3 unformed bowel movements/24h or return to baseline bowel habit 2 weeks after final Fecal Microbiota Transplant (FMT)
Time Frame: 2 weeks after final Fecal Microbiota Transplant (FMT)
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Transplant With Fidaxomicin
Number analyzed (Participants) | 4
Participants | 4

2. Secondary Outcome: Sustained C Difficile Infection (CDI) Resolution (Eight Weeks After Final After Final Fecal Microbiota Transplant (FMT))
Description: Sustained C difficile infection (CDI) resolution defined as lack of C difficile infection (CDI) recurrence 8 weeks after final Fecal Microbiota Transplant (FMT)
Time Frame: 8 weeks after final Fecal Microbiota Transplant (FMT)
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Transplant With Fidaxomicin
Number analyzed (Participants) | 4
Participants | 3

3. Secondary Outcome: Death
Description: Reported death
Time Frame: 8 weeks after final Fecal Microbiota Transplant (FMT); up to 96 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Transplant With Fidaxomicin
Number analyzed (Participants) | 4
Participants | 0

4. Secondary Outcome: Perforation
Description: Colonic perforation
Time Frame: 8 weeks after final Fecal Microbiota Transplant (FMT); up to 96 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Transplant With Fidaxomicin
Number analyzed (Participants) | 4
Participants | 0

5. Secondary Outcome: Infection
Description: Proven infection related final Fecal Microbiota Transplant (FMT)
Time Frame: 8 weeks after final Fecal Microbiota Transplant (FMT); up to 96 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Transplant With Fidaxomicin
Number analyzed (Participants) | 4
Participants | 0

6. Secondary Outcome: Hospitalization
Description: Hospitalization due to C. difficile infection (CDI)
Time Frame: 8 weeks after final Fecal Microbiota Transplant (FMT); up to 96 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Transplant With Fidaxomicin
Number analyzed (Participants) | 4
Participants | 0

7. Secondary Outcome: Colectomy
Description: Surgical Intervention - Colectomy
Time Frame: 8 weeks after final Fecal Microbiota Transplant (FMT); up to 96 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Transplant With Fidaxomicin
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: 8 weeks after final Fecal Microbiota Transplant (FMT); up to 96 days.
Arm/Group | Fecal Transplant With Fidaxomicin
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT03760484/Prot_003.pdf
  • Informed Consent Form (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT03760484/ICF_002.pdf